CLINICAL TRIAL: NCT04965558
Title: Clinical Features and Outcome in Patients With Osseomuscular Type of Wilson's Disease
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: WD-osseomuscular type
Record Dates: First submitted 2021-07-05; First posted 2021-07-16 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Clinical Features and Outcome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The investigators aimed to observe the clinical features and outcome in patients with osseomuscular type of Wilson's disease from a large cohort during long-term follow-up

ELIGIBILITY:
Inclusion Criteria:

* genetically diagnosed WD patients

Exclusion Criteria:

* Deny follow-up

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with wilson disease
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2004-01-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Serum ceruloplasmin | From 2004 through 2030
  Serum ceruloplasmin levels were collected among patients with wilson disease. After confirming a non-Gaussian distribution, the reference range of serum ceruloplasmin level was determined.
Urinary Copper Excretion | From 2004 through 2030
  The measurement of 24-hour urine copper excretions were collected and measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China